CLINICAL TRIAL: NCT03773224
Title: A Randomized Trial on Wound Irrigation in Prevention of Surgical Site Infection After Appendectomy
Brief Title: Role of Wound Irrigation After Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura67
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigation (Active Comparator): Layer by layer irrigation of the surgical wound with gentamicin-saline solution
  Interventions: Procedure: Irrigation
- Control (No Intervention): The surgical wound is closed layer by layer without irrigation

INTERVENTIONS:
Procedure: Irrigation — upon closure of the peritoneum gentamicin-saline solution (160 mg of gentamicin in 400 ml of normal saline 0.9%) will be used for irrigation of every layer of the wound before its closure
  Arms: Irrigation

SUMMARY:
Surgical site infection is a common problem after open appendectomy. Irrigation of the surgical wound by topical antibiotics has been devised as a measure to reduce the incidence of wound infection. The present trial aims to assess the efficacy of layer-by-layer wound irrigation with gentamicin-saline solution in prevention of superficial surgical site infection after open appendectomy for acute uncomplicated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders aging between 18 and 65 years who present with acute appendicitis.
* Patients with perforated appendicitis will be also included.

Exclusion Criteria:

* Patients with appendicular mass, appendicular abscess, generalized peritonitis.
* Patients with other causes of acute abdomen as revealed intraoperatively.
* Patients taking long course of steroid therapy or immunosuppressive treatment,
* Patients unwilling to participate in the trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 2 months after surgery
  The incidence of superficial site infection as detected by clinical examination on follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, Study Chair — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided